CLINICAL TRIAL: NCT02333513
Title: A Study to Evaluate the Safety and Effectiveness of PCV Chemotherapy in Patients With Recurrent High-grade Glioma With IDH1/2 Mutation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Yanda Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YDCR-2014-006; ChiCTR-OOC-15005759 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Recurrent High-grade Glioma
MeSH Terms: conditions — Glioma | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- case group (Experimental)
  Interventions: Drug: Lomustine/Vincristine/Procarbazine

INTERVENTIONS:
Drug: Lomustine/Vincristine/Procarbazine

SUMMARY:
This trial is aimed at evaluating the safety and effectiveness of PCV chemotherapy in patients with recurrent high-grade glioma with IDH1/2 mutation.

DETAILED DESCRIPTION:
This trial is aimed at evaluating the safety and effectiveness of PCV chemotherapy in patients with recurrent high-grade glioma with IDH1/2 mutation. And, this trial is approved by medical ethics committee of hebei yanda hospital. Also, the trial has got a registry code "ChiCTR-OOC-15005759" in China clinical trial registry. Researchers will conduct thsi trial from 2015/02 to 2017/12, and 100 recurrent high-grade glioma with IDH1/2 mutation patients will be recruited. Patients who are recruited will get PCV chemotherapy in ether Hebei Yanda Hospital or Beijing Tiantan hospital, and get follow-ups from clinicians.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of high-grade glioma was established by pathological method,and the recurrency of the disease is ongoing.
* The report of the pathological diagnosis contained the status of IDH gene, and showed that IDH1/2 mutation existed.
* The age of the patient is between 18 years old and 70 years old.
* The condition of the patient permits the procedure of chemotherapy using PCV schema.
* The patient is informed consent, and willing to join in this research.

Exclusion Criteria:

* The diagnosis is not recurrent high-grade glioma.
* The diagnosis of high-grade glioma was not established by pathological method.
* No molecular neuropathological report is available, or the report showed that IDH1/2 mutation did not exist.
* The age of the patient does not meet the requirement of this research.
* The condition of the patient does not permit the procedure of chemotherapy using PCV schema.
* There are other conditions that the clinicians believe that the PCV chemotherapy is not appropriate for the patient.
* The patient is not willing to join in this research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 12 months or later

SECONDARY OUTCOMES:
6-month progression-free survival rate | 6 month
12-month progression-free survival rate | 12 month
6-month survival rate | 6 month
12-month survival rate | 12 month
6-month life quality as measured by European Organization for the Research and Treatment of Cancer Quality of Life questionnaires(EORTC QLQ-C30,EORTC QLQ-BN20) and other methods | 6 month
12-month life quality as measured by European Organization for the Research and Treatment of Cancer Quality of Life questionnaires(EORTC QLQ-C30,EORTC QLQ-BN20) and other methods | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ji, Medical Doctor, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Hebei Yanda Hospital, Sanhe, Hebei